CLINICAL TRIAL: NCT01983631
Title: The Effect of Whole Body Vibration Training on Neuromuscular Property in Individuals With Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Associate Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-1184B
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Spinocerebellar Ataxia
Keywords: Whole body vibration; Reciprocal inhibition; Spinocerebellar ataxia; voluntary activation level
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- WBV group (Experimental): Stage 1: Short-term Whole body vibration(3 minutes in half-squatting position)
  Interventions: Other: Whole body vibration training
- Non-WBV group (No Intervention): Stage 1 : Controlled group
- training group (Experimental): Stage 2: Long-term WBV training (3 sessions per week for 4 weeks)
  Interventions: Other: Whole body vibration training
- non-training group (No Intervention): Stage 2: Controlled group

INTERVENTIONS:
Other: Whole body vibration training
  Arms: WBV group; training group

SUMMARY:
The Cerebellum contains ten percent of the total volume of the brain and receives brain, spinal cord and vestibular sensory input. The organization of vestibular and somato-sensory afferent informations are also reported to be impaired in patients with cerebellum dysfunctions. Ataxia and impaired balance control are common symptoms in individuals with spinocerebellar ataxia (SCA). Previous studies have shown that patient with cerebellar damage are usually agonist and antagonist muscle coordination problem. Past studies also found the regulation of reciprocal Ia inhibition was impaired in patients with spinaocerebellar ataxia. In chronic phase, weakness might be developed due to deconditioned. All deficits mentioned above might lead to a decrease functional ability. Therefore, increasing somato-sensory and vestibular input, normalizing the modulation of recriprocal inhibition, and improve muscle strength might be able to improve the functional abilities of individuals with SCA.

Recently, whole body vibration (WBV) has been trained for health groups. Studies showed that WBV training were able to improve muscle strength, balance control, and functional ability. However, there is no evidence showed that whether the whole body vibration training can affect the brain and spinal cord for the regulation of neural circuits. Whether also can affect for maximal voluntary contraction and improve central fatigue. No previous studies that whole body vibration training for SCA.

Therefore, the purpose of this research was to investigate the intracortical facilitation and inhibition, reciprocal Ia inhibition, low frequency depression, maximal voluntary contraction, interpolated twitch technique to compare the different between the SCA and health subject. Also to investigate the short term and long term effect of WBV.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinocerebellar ataxia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Muscle twitch force | Baseline, 4 weeks.
  Measure of changes in muscle twitch force by interpolation twitch technique
Muscle voluntary activity level | Baseline, 4 weeks
  Measure of changes in muscle voluntary activity level by interpolation twitch technique.
Balance | Baseline, 4 weeks
  Measure of changes in berge balance scale and one-leg standing.
Severity of cerebellar ataxia | Baseline, 4 weeks
  Measure of changes in international cooperative ataxia rating scale(ICARS).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan